CLINICAL TRIAL: NCT00640380
Title: A Comparison Between Neurostimulation and Loss of Resistance for Cervical Paravertebral Blocks
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: De QH Tran, Anesthesia Department
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: GEN-07-052
Record Dates: First submitted 2008-03-17; First posted 2008-03-21 (Estimated); Last update posted 2008-04-11 (Estimated); Status verified 2008-04

CONDITIONS: Shoulder Surgery
Keywords: cervical; paravertebral; block
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): CPVB with NS
  Interventions: Other: Nerve stimulation
- 2 (Active Comparator): CPVB with LOR
  Interventions: Other: Loss of resistance to air

INTERVENTIONS:
Other: Nerve stimulation — CPVB with NS
  Arms: 1
Other: Loss of resistance to air — CPVB with LOR
  Arms: 2

SUMMARY:
Cervical paravertebral blocks (CPVBs) target the brachial plexus from a puncture site situated in the posterior aspect of the neck and represent an alternative to interscalene blocks (ISBs) for shoulder and proximal humeral surgery. Randomized controlled trials comparing CPVB and ISB have found no significant differences in success rate, onset and offset times. Because of the reliability of their cutaneous landmarks, CPVBs have become part of the investigators' standard practice. With this approach, the brachial approach can be identified either with loss of resistance to air (LOR) or nerve stimulation (NS). While some authors have used only LOR and reported good success rates, others have hypothesized that NS may increase the reliability of the block. In the proposed study, for the first time, the 2 methods will be formally compared.

ELIGIBILITY:
Inclusion Criteria are:

* age between 18 and 70 years
* American Society of Anesthesiologists classification 1-3
* body mass index between 20 and 28

Exclusion criteria are:

* adults who are unable to give their own consent
* pre-existing obstructive or restrictive lung disease (assessed by history and physical examination)
* pre-existing neuropathy (assessed by history and physical examination)
* coagulopathy (assessed by history and physical examination and, if deemed clinically necessary, by blood work up ie platelets≤ 100, International Normalized Ratio≥ 1.4 or prothrombin time ≥ 50)
* renal failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up ie creatinine≥ 100)
* hepatic failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up ie transaminases≥ 100)
* allergy to local anesthetic agents (LA)
* pregnancy
* prior cervical spine surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2008-05; Primary Completion 2008-10 (Estimated); Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
Success | 8 months

SECONDARY OUTCOMES:
performance time, onset time, side effects | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: De QH Tran, MD, FRCPC, Principal Investigator — McGill University
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada